CLINICAL TRIAL: NCT01095913
Title: Near-Infrared Imaging of Fluorescent Dyes for Lymph Node Mapping
Brief Title: Fluorescent Dyes for Lymph Node Mapping
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other); National Cancer Institute (NCI) (NIH); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0564
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer
Keywords: Near-Infrared Imaging; Fluorescent Dyes; Lymph Node Mapping; Indocyanine green; IC-Green; nonradioactive optical imaging; fluorescent contrast agent; ICG; lymph nodes; axillary nodal dissection
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IC-Green Injections (Experimental): ICG Injections performed after induction of anesthesia for surgery; 25 µg ICG/injection, with injections of 0.1 cc each to be made starting in the hand, arm, and areolar regions of the breast.
  Interventions: Drug: Indocyanine green (ICG)

INTERVENTIONS:
Drug: Indocyanine green (ICG) — Injections performed after induction of anesthesia for surgery; 25 µg ICG/injection, with injections of 0.1 cc each to be made starting in the hand, arm, and areolar regions of the breast.
  Other Names: IC-Green

SUMMARY:
The goal of this clinical research study is to find lymph nodes before surgery using a dye called indocyanine green (IC-Green).

Objectives:

1. To determine the feasibility of using nonradioactive optical imaging techniques with indocyanine green (ICG) as a fluorescent contrast agent to identify all axillary lymph nodes.
2. To determine the feasibility of using nonradioactive optical imaging techniques with ICG as a fluorescent contrast agent to characterize lymphatic architecture and function in women with breast cancer who are scheduled for axillary node dissection.

DETAILED DESCRIPTION:
IC-Green Injections:

If you are found to be eligible to take part in this study, a member of the study staff will give you between 6-16 injections of IC-Green through a needle in your hand, arm, and breast. The study doctor will discuss the number of injections that you will receive in more detail. The injections will be given after you are under anesthesia.

These IC-Green injections will allow researchers to see the flow of the liquid through your body during imaging and locate the lymph nodes that will be removed during your standard of care surgery. After all of the IC-Green injections have been given, the imaging procedure will begin. Researchers will use an experimental camera that shines a special red light onto your skin causing the IC-Green to glow when the images are taken. The red light is like the red light in a grocery store scanner. The imaging procedure will take about 1 hour to complete.

Before the IC-Green injections and during imaging, a member of the research staff will monitor and record your vital signs (blood pressure, breathing rate, heart rate, and temperature).

After the IC-Green injections, a study staff member will closely monitor the injection site for possible side effects every 15 minutes during the first hour, and then every 30 minutes during the second hour. A study staff member will call you the next day and ask you to take your temperature. This phone call should last about 5 minutes.

Follow-Up Evaluation:

If you spend the night in the hospital after your surgery, a study staff member will visit you for a follow-up the day after surgery. At this visit, your temperature will be recorded and you will be asked how you are feeling and if you have had any side effects. The visit should last about 10 minutes.

If you do not spend the night in the hospital after surgery, you will be contacted by phone the day after surgery. You will be asked the same questions described above, as well as what your temperature is. The phone call should last about 10 minutes.

Length of Study:

After all of the images have been taken, and the follow-up evaluation is complete, your participation in this study will be over.

This is an investigational study. IC-Green is FDA approved and commercially available for mapping heart, liver, and eye function. The use of IC-Green for mapping the lymph nodes in breast cancer patients is investigational.

The experimental camera, and the images taken with it, are being used for research purposes only and will not be used to manage your treatment.

Up to 20 patients will be take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years of age or older
2. Diagnosis of breast cancer requiring axillary nodal dissection
3. Negative urine pregnancy test within 72 hours prior to study drug administration, if female of childbearing potential
4. Females of childbearing potential who agree to use a medically accepted method of contraception for a period of one month following the study. Medically acceptable contraceptives include (i) hormonal contraceptives (such as birth control pills, Depo-Provera, or Lupron Depot) if such use is approved by the subject's Oncologist; (ii) barrier methods (such as a condom or diaphragm) used with a spermicide, or (iii) an intrauterine device (IUD).
5. Continuation of Inclusion #4: Non-childbearing potential is defined as physiologically incapable of becoming pregnant, including any female who is post-menopausal; postmenopausal is defined as the time after which a woman has experienced 12 consecutive months of amenorrhea (lack of menstruation).
6. Patients with a positive fine needle aspirate or core biopsy of their axillary nodes

Exclusion Criteria:

1. Women who are pregnant or breast-feeding
2. Persons who are allergic to iodine
3. A female of child-bearing potential who does not agree to use an approved contraceptive for one month after study participation
4. History of ipsilateral axillary surgery including sentinel node biopsy
5. Any patient who does not meet inclusion criteria for study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Nodes Identified by ICG Among All Resected Lymph Nodes for Each Patient | Injection and Imaging procedure takes 1+ hour to complete

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, MD, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of Texas Health Science Center - Houston, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center website — http://www.mdanderson.org